CLINICAL TRIAL: NCT06306963
Title: Prevalence of Gastric Motor Dysfunction and Upper GI Symptoms in Gastric Antral Vascular Ectasias
Acronym: GAVE
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Cairn Diagnostics (Industry)
Responsible Party: Principal Investigator, Xiao Jing (Iris) Wang, Principal Investigator, Mayo Clinic
Other Study IDs: 23-004669
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Gastric Antral Vascular Ectasia; Cirrhosis; Chronic Kidney Disease
MeSH Terms: conditions — Gastric Antral Vascular Ectasia; Fibrosis; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cirrhosis or Chronic Kidney Disease With Gastric Antral Vascular Ectasia: Patients with Gastric Antral Vascular Ectasia with cirrhosis or chronic kidney disease will undergo a gastric emptying breath test. This test is designed to show how quickly the stomach empties solids by measuring labeled carbon dioxide in a patient's breath.
  Interventions: Diagnostic Test: Gastric Emptying Breath Test
- Cirrhosis or Chronic Kidney Disease Without Gastric Antral Vascular Ectasia: Patients without Gastric Antral Vascular Ectasia with cirrhosis or chronic kidney disease will undergo a gastric emptying breath test. This test is designed to show how quickly the stomach empties solids by measuring labeled carbon dioxide in a patient's breath.
  Interventions: Diagnostic Test: Gastric Emptying Breath Test

INTERVENTIONS:
Diagnostic Test: Gastric Emptying Breath Test — 13C-Spirulina GEBT (Cairn Diagnostics) is non-radioactive, non-invasive breath based test validated against scintigraphy for the measurement of gastric emptying. Patients will be mailed test kits to be done in their homes remotely along with telehealth assistance from the study team. After overnight fast and providing duplicate pre-meal breath samples, the patient consumes 27 grams of re-hydrated, precisely formulated, pasteurized scrambled egg mix containing a dose of 43 mg of 13C (provided by approximately 100 mg of 13C-Spirulina), 6 saltine crackers and 6 ounces (180 mL) of potable water. The caloric value of the meal is approximately 230 kCal.Patient will provide breath samples into provided glass tubes before and after test meal administration which are then mailed back to a central laboratory for analysis by gas isotope ratio mass spectrometry.
  Other Names: Gastric motor function testing

SUMMARY:
The researchers are trying to find out more about Gastric Antral Vascular Ectasia (GAVE). This is a condition that affects the blood vessels in the stomach, leading to their enlargement and possible bleeding. It can also cause symptoms such as abdominal pain and nausea. By participating in this study, you will help us learn how often these symptoms occur and how they relate to stomach functioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age with endoscopic evidence of Gastric Antral Vascular Ectasia.
* Willingness to participate in the study
* Capacity to provide informed consent.
* No evidence of organic, systemic, or metabolic disease (e.g. diabetes mellitus) to explain the symptoms on routine investigations

Exclusion Criteria:

* Patients with transfusion dependent blood loss.
* Patients with severe decompensated liver disease.
* Patients with end stage renal disease.
* Presence of other diseases (structural or metabolic) which could interfere with interpretation of the study results.
* Pregnant or lactating women.
* Patients who have not had a CBC and differential blood draw completed within the last six months.
* Current heavy alcohol use.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone an endoscopy and found to have GAVE will be included. Patients with underlying cirrhosis or chronic kidney disease and GAVE in comparison to control patients with cirrhosis or chronic kidney disease and no GAVE.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Nepean Dyspepsia Index | baseline
  The Nepean Dyspepsia Index is a 10-item questionnaire that measures dyspepsia problems. Each item is scored from 1-5. 1 = Not at all, 5 = Extremely. Total scores range from 10 - 50, lower scores indicate less dyspepsia problems, higher scores indicate more dyspepsia problems.
Abridged Bowel Disease Questionnaire | baseline
  The Abridged Bowel Disease Questionnaire is a 16-item questionnaire that measures Bowel Disease symptoms. Each item is scored as yes or no. Scores answering yes indicate more bowel disease, and scores answering no indicate less or no bowel disease.
Leuven Postprandial Distress Scale | baseline
  The Leuven Postprandial Distress Scale is an 8-item questionnaire that measures symptoms of dyspepsia. Each item is scored from 1-5. 1 = Absent, 5 = very severe. Total scores range from 0-40 Lower scores indicate less or no symptoms of dyspepsia, higher scores indicate more symptoms of dyspepsia.

SECONDARY OUTCOMES:
GEBT Breath Test | 6 Hours
  The C-Spirulina Gastric Emptying Breath Test is a non-radioactive, Non-invasive test for measurement of the rate in gastric emptying in adults by measuring the C-13 levels in the breath.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Jing Wang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szarka LA, Camilleri M, Vella A, Burton D, Baxter K, Simonson J, Zinsmeister AR. A stable isotope breath test with a standard meal for abnormal gastric emptying of solids in the clinic and in research. Clin Gastroenterol Hepatol. 2008 Jun;6(6):635-643.e1. doi: 10.1016/j.cgh.2008.01.009. Epub 2008 Apr 14. PMID 18406670
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials